CLINICAL TRIAL: NCT00590473
Title: Sacral Neuromodulation: Bilateral Placement vs. Unilateral Placement in Patients With Interstitial Cystitis
Brief Title: Sacral Neuromodulation in Patients With IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71692
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial Cystitis; IC; Neuromodulation; Interstim Therapy
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Unilateral Placement of Interstim IPG
  Interventions: Device: Interstim
- 2 (Active Comparator): Bilateral Placement of Interstim IPG
  Interventions: Device: Interstim

INTERVENTIONS:
Device: Interstim — Unilateral vs. Bilateral Placement of Interstim IPG

SUMMARY:
The hypothesis for this study is that bilateral sacral neuromodulation will improve symptoms of interstitial cystitis by at least 25% when compared to unilateral sacral neuromodulation as reported by patient's responses to the Interstitial Cystitis Symptom and Problem Indices.

This study will be a prospective randomized study comparing bilateral to unilateral sacral neuromodulation. The study population will include all patients diagnosed with interstitial cystitis, using the NIDDK criteria, having staged sacral neuromodulator stimulators placed at Hahnemann University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of interstitial cystitis for at least 6 months.
* At least 18yrs old and less than 80.
* Symptoms of urgency (>4 on the visual analog scale).
* Symptoms of urinary frequency (>8 episodes/day as recorded on a voiding diary)
* Symptoms of pelvic pain (>4 on the visual analog scale for pelvic pain).
* Interstitial Cystitis refractory to more conservative treatments such as behavioral modification, dietary intervention, or medical therapy for at least 6 months.
* Able to make medical decisions for herself.
* Presence of either glomerulations of Hunner's ulcer on cystoscopic examination.
* Participant must agree to use a medically acceptable method of contraception throughout the entire study period, and for 7 days after the study period. Medically acceptable methods of contraception include abstinence, birth control pills or patches, diaphragm with spermicide, IUD, condom with vaginal spermicide, surgical sterilization, post menopausal for at least 1 year, implants or injections, or vasectomized partner.
* Must give written informed consent to participate in this study.

Exclusion Criteria:

* Prior sacral neuromodulation.
* Participant is currently pregnant or breastfeeding.
* Male.
* Urinary retention (defined by post void residual greater than 100cc).
* Neurologic deficit.
* Need for future MRI surveillance.
* Involved in any study within the past thirty days or currently enrolled.
* Presence of bladder or ureteral calculi.
* Active genital herpes.
* Uterine, cervical, vaginal, or urethral cancer.
* Urethral diverticulum.
* Cyclophosphamide cystitis.
* Vaginitis.
* Tuberculous cystitis.
* Foreign body within the bladder (indwelling catheter- foley or suprapubic tube, or ureteral stent).
* An employee or a relative of an employee of Medtronic Inc. or The Pelvic and Sexual Health Institute.
* Bladder capacity greater than 350 cc while awake during cystometrogram.
* Duration of symptoms of less than 6 months.
* Detrusor overactivity on cystometrogram.
* Absence of nocturia, defined by greater than 2 voids per sleeping hours.
* Urinary symptoms relieved by either antimicrobials, antiseptics, anticholinergics, or antispasmodics.
* Urinary frequency of less than 8 voids per day.
* Diagnosis of bacterial cystitis or prostatitis within the past 3 months.
* Radiation cystitis.
* Benign or malignant bladder tumors.
* Age less than 18 or greater than 79.
* Participant is currently receiving or has received pelvic radiation.
* Participant is diagnosed with cancer within the past 5 years prior to the start of the study.
* Participant has a history of alcohol or substance abuse within the past 5 years prior to the start of the study.
* Severe or uncontrolled diabetes or diabetes with peripheral nerve involvement.
* Patients with implanted electrical devices (cardiac pacemakers or defibrillators).
* Patients on anticoagulation therapy.
* Planned future exposure to diathermy, microwave, or RF energy.

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To determine if bilateral sacral neuromodulation will reduce the patient's score on the Interstitial Cystitis Symptom and Problem Questionnaire by at least 25% when compared to unilateral sacral neuromodulation in patients with interstitial cystitis. | Post-op, at 6 weeks and at 3 months post-surgery

SECONDARY OUTCOMES:
To determine if bilateral sacral neuromodulation will improve the patient's voiding diary defined as reduction in urinary frequency by 25% from baseline when compared to unilateral sacral neuromodulation in patients with interstitial cystitis | Post-op, at 6 weeks and 3 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kristene E. Whitmore, M.D., Principal Investigator — Drexel University College of Medicine
Locations (1):
- Pelvic and Sexual Health Institute, Philadelphia, Pennsylvania, United States